CLINICAL TRIAL: NCT05053555
Title: High Dose-Rate Brachytherapy for the Treatment of Both Primary and Secondary Unresectable Liver Malignancies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-1255; NCI-2021-09408 (Other: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2021-08-24; First posted 2021-09-22 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Liver Malignant Tumors; Cholangiocarcinoma Metastatic; Pancreatic Cancer; Melanoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Pancreatic Neoplasms; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Prospective cohort ) (Experimental): 20 patients, will undergo initial diagnostic workup, staging and treatment per institutional standard of care. Intervention: High dose rate brachytherapy (HDRBT)
  Interventions: Device: high dose rate brachytherapy
- Group B( Retrospective chart review ) (Experimental): 40 patients who meet same eligibility criteria, but did not receive HDRBT between 1/1/2000 and 1/1/2021.
  Interventions: Device: high dose rate brachytherapy

INTERVENTIONS:
Device: high dose rate brachytherapy — diagnostic workup, staging, and treatment per the institution standard of care
  Arms: Group A (Prospective cohort )
Device: high dose rate brachytherapy — reviewing historical patients who meet the above criteria for group A but did not receive HDRBT between 01/01/2000 and 1/01/2021
  Arms: Group B( Retrospective chart review )

SUMMARY:
Over the past three decades, the treatment of both primary and secondary liver malignancies has been improved by the development and optimization of multiple minimally invasive thermal ablative therapies. These advances have resulted in a myriad of benefits for patients including decreased morbidity, mortality, as well as increased longevity and quality of life. However, these therapies can only be performed within certain parameters. Thermal ablative techniques such as radiofrequency ablation (RFA) and microwave ablation (MVA) are recommended for small lesions under 3 cm due to decreased efficacy when attempting to treat larger lesions. Additionally, large vessels in close proximity to a target lesion may result in heat dissipation, termed the "heat sink" effect, and result in incomplete ablation of the lesion. Furthermore, thermal ablative techniques cause off-target damage when utilized near sensitive structures such as the diaphragm, stomach, or bowel, and if performed near thermosensitive bile ducts, can result in cholestasis . Noting these limitations, percutaneous high-dose-rate brachytherapy was brought into clinical practice by Ricke et al. in Europe in 2002 . This therapy utilizes an iridium-192 (192Ir) isotope to administer a cytotoxic dose of radiation to a target lesion. It is not susceptible to heat sink effects and can also deliver radiation with the precision necessary to cause tumor death without destroying the integrity of neighboring structures. Additionally, it can be used to treat larger tumors (>3cm) as it is not associated the same size limitations as ablative techniques and can also be utilized to treat lesions that are not amenable to intra-arterial therapies (such as trans-arterial chemoembolization and yttrium-90 radioembolization).

Since its inception, HDRBT has been evaluated through multiple studies investigating its use to treat lesions throughout the body including both primary and secondary liver malignancies such as hepatocellular carcinoma (HCC), cholangiocarcinoma, metastasis to the liver from colorectal cancer, pancreatic cancer , melanoma , and breast cancer . Its use in treating lymph node metastases has also been investigated . These studies have demonstrated the feasibility, safety, and clinical effectiveness of this method, establishing it as a therapeutic option when use of thermal ablation therapies is restricted. Most studies however, have been retrospective and have been performed outside the United States.

Studying this therapy will add a crucial treatment option to our current armamentarium, filling a gap in currently available therapies and additionally allowing for further investigation of the use of HDRBT in a larger and more diverse population.

DETAILED DESCRIPTION:
Primary Objective

-To prospectively evaluate the clinical effectiveness of the use of high dose rate brachytherapy (HDRBT) for the treatment of both primary and secondary unresectable liver malignancies assessed by comparing local tumor control (LTC) rates at 6 months with a historical cohort.

Secondary Objectives

* To compare local tumor control rates at 3-month intervals between cohorts for the duration of the study (3 months, 9 months, 12 months, etc.).
* To compare overall survival (OS) and progression-free survival (PFS) between cohorts.

ELIGIBILITY:
Inclusion Criteria:

* GROUP A: Patients with liver lesions must be over the age of 18
* GROUP A: Any patient with up to five unresectable tumors that are:

  * At least 3 cm (largest diameter in the axial plane)
  * In close proximity to large blood vessels
  * In close proximity to sensitive structures (bowel, stomach, diaphragm, liver capsule, liver hilum, bile ducts)
  * Associated with difficult endovascular access to one or more feeding arterial branches (hypovascular tumors)
  * Associated with a large shunt fraction to other vital organs
* GROUP B: Historical patients who meet the above criteria for group A but did not receive HDRBT between 01/01/2000 and 1/01/2021

Exclusion criteria:

* Active infectious disease
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, interstitial lung disease, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with polymetastatic disease with the exception of those patients who may benefit from therapy addressing local complications directly related to the target lesion diminishing quality of life such as pain, vascular/biliary occlusion, and liver disfunction
* Pregnancy (sexually active patients must be on birth control while participating in this study)
* Child-Pugh class C
* Total serum bilirubin > 2 mg/dl
* Platelet count < 50,000/ul
* International normalized ratio (INR) > 1.5

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-04-24 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
To prospectively evaluate the clinical effectiveness of the use of high dose rate brachytherapy (HDRBT) for the treatment of both primary liver malignancies. | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Kuban, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org